CLINICAL TRIAL: NCT04459351
Title: PHenotyping patiENts Admitted to Hospital With cOvid-19 Infection and idenTifYing Prognostic markErs
Acronym: PHENOTYPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W20/035
Record Dates: First submitted 2020-06-18; First posted 2020-07-07 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus; Corona Virus Infection; COVID-19; 2019nCoV; 2019 Novel Coronavirus Infection
Keywords: COVID-19; Blood phenotyping
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * Blood samples: 20 additional mls taken at each routine follow-up visit.
  * Endobronchial samples (washings/brushings/biopsy) if a bronchoscopy is deemed necessary for the clinical care of the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PHENOTYPE is an investigator-led, observational cohort study which aims to explore the long-term outcomes of patients with COVID-19 infection and to identify potential risk factors and biomarkers that can prognosticate disease severity and trajectory.

DETAILED DESCRIPTION:
In 2019, a novel coronavirus, SARS-CoV-2 was first identified in Wuhan, China. SARS-CoV-2 infection, denominated COVID-19, causes a predominantly respiratory illness, which varies from mild respiratory symptoms to multi-organ failure and death. In March 2020, COVID-19 was designated pandemic status and as of May 2020 there have been more than 3.7 million cases reported worldwide and 257,000 deaths attributed. In the UK, COVID-19 has caused more than 30,000 deaths to date.

Although respiratory symptoms are the commonest presentation, numerous systemic complications of COVID-19 have been identified, including those affecting the cardiovascular, neurological, gastroenterological, and renal systems. The long-term impact of these complications on survivors and the risk factors for long term sequelae is not presently known. It is likely that increased frailty and psychological sequelae will be significant, which could lead to a persistent reduction in quality of life, as observed in the previous SARS pandemic.

This cohort study aims to evaluate the respiratory, cardiac, renal and psychological outcomes of patients diagnosed with COVID-19 infection and determine the pathophysiological mechanisms that contribute to disease severity and disease burden.

ELIGIBILITY:
Inclusion Criteria

* Aged 18 years or older
* Confirmed COVID-19 infection (as per national guidelines)
* Attending follow-up outpatient visit post hospital attendance with COVID-19 infection

Exclusion Criteria

There are no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged 18 or older) who have attended hospital with proven COVID-19 infection and are being followed up in clinic are potential candidates for study enrolment. A member of the clinical or research team will screen the patient against the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Identification of baseline characteristics which correlate with disease severity | Based on clinical need - Up to 1 year follow up.
  The primary purpose is to characterise the different presentations and features of COVID-19 and outcomes.
Identification of blood biomarkers which correlate with disease severity | Based on clinical need - Up to 1 year follow up.
  Relationship between changes in markers of inflammation (CRP, D dimer, ferritin, fibrinogen, pro-calcitonin) and pulmonary, renal and cardiac complications post hospitalisation for Covid-19 infection.
Genomic analysis of blood samples to look for genetic susceptibility to severe disease presentations | Based on clinical need - Up to 1 year follow up.
  Genomic, proteomic and transcriptomic analysis of blood samples to look for genetic susceptibility to severe disease presentations and to identify new biomarkers that predict disease severity or disease trajectory

SECONDARY OUTCOMES:
Incidence | Based on clinical need - Up to 1 year follow up.
  Incidence of:
  * Interstitial lung disease
  * Pulmonary embolism
  * Pulmonary hypertension as determined by pulmonary artery systolic pressure on echocardiogram or mean pulmonary artery pressure on right heart catheterisation if performed
  * Renal dysfunction (as defined by new persistent impairment of egfr or new sustained protenuria measured using urinary protein-creatinine ratio)
  * Cardiac dysfunction (new LV or RV systolic dysfunction on echocardiogram)
  * Psychological distress as measured using Hospital anxiety and depression scale
Change in respiratory symptom scores | Based on clinical need - Up to 1 year follow up.
  Assessed through Leicester Cough Questionnaire: Domain scores 1-7; Total scores 3-21
Change in respiratory symptom scores | Based on clinical need - Up to 1 year follow up.
  Assessed through the modified Medical Research Council Dyspnoea Scale: Scores range from 0-4.
Change in frailty and quality of life scores | Based on clinical need - Up to 1 year follow up.
  Assessed thought the Short Form Survey (36): 8 scales, each scored between 0-100.
Change in frailty and quality of life scores | Based on clinical need - Up to 1 year follow up.
  Assessed through the Clinical Frailty Scale: Scores range from 1-9.
Relationship between serum markers and clinical outcomes | Based on clinical need - Up to 1 year follow up.
  D dimer/ fibrinogen and new pulmonary embolism
Relationship between serum markers and clinical outcomes | Based on clinical need - Up to 1 year follow up.
  Troponin/ BNP and cardiac disease
Relationship between serum markers and clinical outcomes | Based on clinical need - Up to 1 year follow up.
  Markers of inflammation (CRP, procalcitonin, ferritin, fibrinogen, D dimer, ESR) and persistent radiological abnormalities

OTHER OUTCOMES:
Thematic analysis of semi-structured interviews exploring the following areas: | Up to 1 year follow up.
  * Changes in health behaviours such as alcohol consumption and tobacco use
  * Mental health and psychological wellbeing
  * Factors affecting compliance with Public Health England guidelines
  * The impact of cultural and religious beliefs on behaviours during the pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MBBS, MD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong, S., Vaughan, A., Quilty-Harper, C. & Liverpool,L. Black people in England and Wales twice as likely to die with covid-19. New Scientist. 2020. Available from: https://www.newscientist.com/article/2237475-covid-19-news-uk-economy-shrank-at-fastest-pace-since-2008/[Accessed: 10th May 2020]
- [Background] Chan KS, Zheng JP, Mok YW, Li YM, Liu YN, Chu CM, Ip MS. SARS: prognosis, outcome and sequelae. Respirology. 2003 Nov;8 Suppl(Suppl 1):S36-40. doi: 10.1046/j.1440-1843.2003.00522.x. PMID 15018132
- [Derived] Vijayakumar B, Tonkin J, Devaraj A, Philip KEJ, Orton CM, Desai SR, Shah PL. CT Lung Abnormalities after COVID-19 at 3 Months and 1 Year after Hospital Discharge. Radiology. 2022 May;303(2):444-454. doi: 10.1148/radiol.2021211746. Epub 2021 Oct 5. PMID 34609195